CLINICAL TRIAL: NCT01137994
Title: A Phase II, Randomized, Open-label Study of Lapatinib Plus Chemotherapy Versus Trastuzumab Plus Chemotherapy as First-line Treatment for Women With HER2-positive and p95HER2-positive Metastatic Breast Cancer
Brief Title: A Phase II, Randomized, Open-label Study of Lapatinib Plus Chemotherapy Versus Trastuzumab Plus Chemotherapy in HER2-positive and p95HER2-positive Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113333
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasms, Breast
Keywords: ErbB2; Trastuzumab; p95HER2; Metastatic Breast Cancer; HER2; Lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Docetaxel; Paclitaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapatinib plus Chemotherapy (Experimental): Lapatinib (1250mg once daily) in combination with chemotherapy (docetaxel, paclitaxel or vinorelbine) selected at the discretion of the investigator
  Interventions: Drug: Lapatinib; Drug: Docetaxel; Drug: Paclitaxel; Drug: Vinorelbine
- Trastuzumab plus Chemotherapy (Experimental): Trastuzumab (either 6mg/kg q3-weekly or 2mg/kg weekly) in combination with chemotherapy (docetaxel, paclitaxel or vinorelbine) selected at the discretion of the investigator
  Interventions: Biological: Trastuzumab; Drug: Docetaxel; Drug: Paclitaxel; Drug: Vinorelbine

INTERVENTIONS:
Drug: Lapatinib — oral, reversible small molecule tyrosine kinase inhibitor of HER2 receptor
  Arms: Lapatinib plus Chemotherapy
Biological: Trastuzumab — monoclonal antibody directed to HER2 receptor
  Arms: Trastuzumab plus Chemotherapy
Drug: Docetaxel — Taxane chemotherapy
Drug: Paclitaxel — Taxane chemotherapy
Drug: Vinorelbine — Vinka alkaloid

SUMMARY:
This is a Phase II, randomized, open-label, multi-center study evaluating the efficacy and safety of lapatinib in combination with chemotherapy versus trastuzumab in combination with chemotherapy in women with HER2-positive and p95HER2-positive metastatic breast cancer (MBC). Eligible subjects will have newly diagnosed metastatic breast cancer (Stage IV) either as a primary diagnosis or as a recurrence following treatment of curative intent; not have received systemic or local treatment for MBC and have breast cancer that is positive for HER2 and p95HER2. The primary objective is to compare progression-free survival (PFS) of lapatinib plus chemotherapy versus trastuzumab plus chemotherapy as first-line treatment in subjects with MBC exhibiting concurrent HER2 overexpression (and/or gene amplification) and expression of carboxy-terminal fragments of HER2 (p95HER2). The secondary objectives are to evaluate overall survival, overall response rate, clinical benefit response rate and the safety as well as tolerability of lapatinib plus chemotherapy and trastuzumab plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years of age
* Histologically or cytologically confirmed invasive breast cancer with distant metastasis(ses) (designated as Stage IV or metastatic breast cancer)

  * Diagnosis with Stage IV or metastatic disease at either primary diagnosis or recurrence
* Not received prior systemic or local treatment (e.g., chemotherapy, endocrine or radiotherapy) for Stage IV/metastatic breast cancer

  * Prior adjuvant and/or neo-adjuvant therapy is permitted
* Documentation of HER2 overexpression or gene amplification, in the invasive component of either a metastatic disease site or primary tumor, defined as: 3+ by IHC and/or HER2/neu gene amplification by fluorescence, chromogenic or silver in situ hybridization [FISH, CISH or SISH; >6 HER2/neu gene copies per nucleus or a FISH, CISH or SISH test ratio (HER2 gene copies to chromosome 17 signals) of ≥2.0]
* Documentation by the central laboratory of positive p95HER2 expression in the invasive component of either a metastatic disease site (preferred) or primary tumor
* No history of CNS metastases (including leptomeningeal involvement) or stable CNS metastases (defined as asymptomatic and off steroids for ≥ 3 months)
* Baseline Left Ventricular Ejection Fraction (LVEF) ≥50% measured by echocardiography (ECHO) or multi-gated acquisition scan (MUGA)
* Recovered or stabilized from all adverse events associated with prior anti-cancer therapies, including radiotherapy, at the time of screening
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Have adequate marrow and organ function as defined as:

SYSTEM LABORATORY VALUES Hematologic ANC ≥1.5 x 109/L Hemoglobin ≥9 g/dL (after transfusion if needed) Platelets ≥100 x 109/L Hepatic Albumin ≥ 2.5 g/dL Serum bilirubin ≤1.5 x ULN unless due to Gilbert's syndrome AST and ALT ≤3 x ULN Renal Calculated creatinine clearance ≥ 40 mL/min Serum Creatinine ≤1.5 mg/dL or 132.6µmol/L (Abbreviations: ANC, absolute neutrophil count; ULN, upper limit of normal; AST, aspartate aminotransferase; ALT, alanine aminotransferase)

* Women of childbearing potential, including women whose last menstrual period was <12 months ago (unless surgically sterile) must have a negative serum pregnancy test and agree to use effective contraception, as defined in protocol
* Signed Informed Consent Form

Exclusion Criteria:

* History of other malignancy. Exception: Subjects who have been disease-free for 5 years or subjects with a history of completely resected non-melanoma skin cancer (basal or squamous) are eligible
* Concurrent anti-cancer treatment or concurrent treatment with an investigational drug
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment
* Prior treatment with anti-HER2 therapy, except trastuzumab or lapatinib (time from last dose of trastuzumab or lapatinib to randomization must be ≥3 months)
* Serious cardiac illness or medical condition including but not confined to:

  * Uncontrolled arrhythmias
  * Uncontrolled or symptomatic angina
  * History of congestive heart failure (CHF)
  * Documented myocardial infarction <6 months from study entry
* Current active hepatic or biliary disease (with exception of Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Concurrent disease or condition, or any pre-existing medical disorder that in the opinion of the investigator may interfere with the subject's safety, obtaining informed consent or compliance to the study procedures
* Pregnant or lactating female
* Any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels (consult with GSK Medical Monitor if uncertain about eligibility)
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study drugs or their excipients that, in the opinion of the investigator contra-indicates participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2016-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Time from randomization to disease progression

SECONDARY OUTCOMES:
Overall Survival | end of study
Overall response rate (ORR: complete response [CR] or partial response [PR]) | end of study
Clinical benefit response rate (CBR: CR or PR at any time, or stable disease [SD] >=24 weeks | end of study
Safety and tolerability of lapatinib plus chemotherapy and trastuzumab plus chemotherapy | end of study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline